CLINICAL TRIAL: NCT02046304
Title: A Phase I Study of Preoperative Concomitant Gemcitabine and External-Beam Radiation Therapy and Surgical Resection for Patients With Extremity and Trunk Soft Tissue Sarcomas
Brief Title: PP-Gemcitabine & External Beam Radiation-Sarcomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-532
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Sarcoma
Keywords: Sarcoma; Soft Tissue Sarcomas; STS; Extremity and Trunk; Gemcitabine; Gemcitabine Hydrochloride; Gemzar; External beam radiation therapy; EBRT; Radiotherapy; XRT
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Radiation Therapy (Experimental): Patients receive concurrent chemoradiation (days 1 - 33) consisting of external beam radiotherapy (EBRT) plus gemcitabine, administered in a phase I dose escalation format until MTD is reached. EBRT delivered preoperatively (for patients with measurable disease) or postoperatively (for patients who have undergone pre-referral excisional biopsy) to a dose of 50 Gy in 25 fractions at 2.0 Gy per fraction. Radiotherapy given once daily (Monday through Friday) for 5 weeks. Surgical resection of the post-treatment tumor mass performed 4 to 8 weeks after the final dose of gemcitabine. Gemcitabine administered intravenously (IV) on days 1, 8, 22, 29, 43, and 50, concurrently with radiotherapy. Starting dose of gemcitabine 400 mg/m2 by vein once a week.
  Interventions: Drug: Gemcitabine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Gemcitabine — Starting dose: 400 mg/m2 by vein on days 1, 8, 22, 29, 43, and 50.
  Other Names: Gemcitabine Hydrochloride; Gemzar
Radiation: Radiation Therapy — Radiation therapy dose of 50 Gy in 25 fractions at 2.0 Gy per fraction. Radiotherapy given once daily (Monday through Friday) for 5 weeks.
  Other Names: XRT; EBRT; Radiotherapy

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of gemcitabine that can be given with radiotherapy before surgery to treat sarcoma. This study will also look at how well this treatment controls sarcoma.

DETAILED DESCRIPTION:
Before the start of treatment, participants will have a physical exam, blood tests, a MRI scan, and a chest x-ray. A PET scan may be done if thought necessary.

Participants will receive the drug gemcitabine by vein along with radiation therapy on Days 1, 8, 22, 29, 43, and 50. Radiation treatments will be given 5 days a week for 5 weeks. The gemcitabine and radiotherapy will be given on an outpatient basis. Chemotherapy and/or radiotherapy may be stopped if side effects become severe.

About 4 to 6 weeks after the final dose of gemcitabine, surgery will be done to remove the tumor or to remove any previous surgical scar and leftover tumor.

During the combined treatment, participants will be seen weekly by the doctor in charge of radiotherapy or by the study nurse. Blood tests will be done every week during treatment. A MRI scan and a chest x-ray will be done within 14 days before surgery. A PET scan will be done if thought necessary.

After the surgery is done, participants will return to M. D. Anderson for follow-up visits every 4 months for the first 2 years, every 6 months for 3 years, and then yearly from then on. An ultrasound and MRI scan (of the extremity or trunk) will be done 3 months after completion of all treatment. Ultrasound scans will be performed at each visit. A MRI scan will only be done again at later visits if needed.

This is an investigational study. Gemcitabine is approved for use by the FDA. Its use together with radiation therapy in this study is experimental. About 36 individuals will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cytologic or histologic proof of Grade II or III resectable soft tissue sarcoma of the extremity or trunk.
2. Patients with both measurable and non-measurable disease. Patients who are S/P pre-referral excision will be eligible.
3. Inclusion of patients with a prior history of malignancy will be at the discretion of the Study Chairman.
4. Patients must have a Zubrod Point Scale of 0 or 1.
5. Absolute neutrophil count must be > 1,500 cells/mm; platelet count greater than or equal to 100,000 platelets/ml; serum creatinine less than or equal to 1.8 mg/dl, serum glutamate oxaloacetate transaminase (SGOT)/serum glutamate pyruvate transaminase (SGPT) less than or equal to 3 x normal, total bilirubin less then or equal to 1.5 mg/dl.
6. Patients must have no uncontrolled coexisting medical conditions.
7. Women of childbearing potential must not be pregnant or breast feeding and must practice adequate contraception.
8. All patients must sign an informed consent.

Exclusion Criteria:

1) Patients with a history of prior radiotherapy in the area of the primary tumor or those in whom the anticipated radiation field would include the perineum, scrotum, or vaginal introitus will not be eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2001-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Preoperative Gemcitabine with External-Beam Radiation Therapy | 6 weeks
  The maximum tolerated dose (MTD) defined as the dose having posterior expected toxicity importance score (TIS) closest to the target 1.65 at the end of the trial.

SECONDARY OUTCOMES:
Response to Preoperative Gemcitabine with External-Beam Radiation Therapy | 3 months after completion of all treatment
  Response to preoperative chemoradiotherapy measured by comparing pre- and post-treatment MRI scans using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Evaluation of the MRI-defined change used to measure radiographic response.

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Pisters, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org